CLINICAL TRIAL: NCT00550628
Title: Pilot Study of Ex-Vivo Molecular Polyp Imaging Using 18-F Fluorodeoxyglucose (FGD) Positron Emission Tomography (PET) in the Determination of Protein and Gene Expression Signatures of Premalignant Polyps
Brief Title: Fludeoxyglucose F 18 PET Imaging in Determining Protein and Gene Expression Signatures in Patients With Premalignant Polyps or Colon Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 07-114; P30CA008748 (NIH); MSKCC-07114
Record Dates: First submitted 2007-10-25; First posted 2007-10-30 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Colorectal Cancer; Neoplasm of Uncertain Malignant Potential
Keywords: neoplasm of uncertain malignant potential; colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — DNA Methylation; In Situ Hybridization, Fluorescence; Gene Expression Profiling; Polymerase Chain Reaction; Reverse Transcriptase Polymerase Chain Reaction; Immunoenzyme Techniques; Immunohistochemistry; Biopsy; Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue

GROUPS / COHORTS (1):
- resection of a non-sarcomatous primary colon neoplasm: The surgically removed colon will undergo ex-vivo imaging after examination in pathology. A PET scanner will be used to acquire a scan of the whole specimen.
  Interventions: Genetic: DNA methylation analysis; Genetic: fluorescence in situ hybridization; Genetic: gene expression analysis; Genetic: polymerase chain reaction; Genetic: protein expression analysis; Genetic: reverse transcriptase-polymerase chain reaction; Other: diagnostic laboratory biomarker analysis; Other: immunoenzyme technique; Other: immunohistochemistry staining method; Procedure: biopsy; Procedure: therapeutic conventional surgery; Radiation: fludeoxyglucose F 18

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: fluorescence in situ hybridization
Genetic: gene expression analysis
Genetic: polymerase chain reaction
Genetic: protein expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: diagnostic laboratory biomarker analysis
Other: immunoenzyme technique
Other: immunohistochemistry staining method
Procedure: biopsy
Procedure: therapeutic conventional surgery
Radiation: fludeoxyglucose F 18

SUMMARY:
RATIONALE: Diagnostic imaging procedures, such as fludeoxyglucose F 18 PET, may be effective in detecting cancer or recurrence of cancer, or premalignant polyps.

PURPOSE: This clinical trial is studying fludeoxyglucose F 18-PET imaging to see how well it works in determining protein and gene expression signatures in patients with premalignant polyps or colon cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the feasibility of ex-vivo imaging of colon cancer and colon polyps using fludeoxyglucose F 18 positron emission tomography (FDG PET).
* To evaluate the differences in molecular and genetic profiles between FDG-positive polyps and FDG-negative polyps to suggest what gene mutations and abnormal mRNA and/or protein expressions may be required for FDG avidity ("signature" for FDG avidity).

Secondary

* To evaluate the differences in molecular and genetic profiles between FDG-positive polyps and FDG-positive cancers to suggest what gene mutations and abnormal mRNA and/or protein expressions may be required for cancer formation ("signature" for cancer).
* To evaluate the differences in molecular and genetic profiles between normal colonic mucosa, polyps, and cancer.
* To evaluate the differences and similarities in molecular and genetic profiles between FDG-positive cancers and polyps.

OUTLINE: Part I: Patients receive fludeoxyglucose F 18 (FDG) IV followed 45-60 minutes later by surgery to remove part or all of the colon. Tissue samples of the colon undergo positron emission tomography (PET) imaging.

Part II: Tissue samples are analyzed for glucose transporters proteins (Glut-1, 2, 3, 4, 5, 7) via IHC; presence of K-ras mutation (invariable mutant site on codon 12, 13) via PCR; 18q deletion via fluorescence in situ hybridization (FISH) or DCC IHC; MCT-1, Hex-1, Hex-2, and COX-2 expression levels via quantitative RT-PCR method or western blot; APC mutation via PCR- In Vitro Synthesized-Protein Assay or RT-PCR direct sequencing method; p53 mutation detection via immunochemistry, RT-PCR direct sequence methods, and western blot; methylation alteration of MGMT, CDKN2A, HLTF, MLH1, TIMP3, HIF1, BNIP3, and HRK via methylation detecting microchip; and specific gene methylations via methylation-specific PCR. Some tissue samples may be saved and banked for future studies.

ELIGIBILITY:
Subject Inclusion Criteria:

* Patients eligible for entry into the study are those:
* Age 15 to 100
* Undergoing resection of a non-sarcomatous primary colon neoplasm who also has 2 or more adenomas each greater than or equal to 7-10mm in size which are anticipated to be removed with the colon specimen.
* It will be known from MSKCC or outside studies (barium enema, endoscopy, PET/CT, or CT colonography) that the patient has at least 2 proven adenomas 7-10 mm or greater and a primary colon neoplasm

Subject Exclusion Criteria:

* Insulin-dependent diabetics (as established by routine history and presurgical laboratory tests).

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: MSK clinic
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2007-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of ex-vivo imaging of colon cancer and colon polyps using fludeoxyglucose F 18 positron emission tomography (FDG PET) | 2 years

SECONDARY OUTCOMES:
Differences in molecular and genetic profiles between FDG-positive polyps and FDG-negative polyps to suggest what gene mutations and abnormal mRNA and/or protein expressions may be required for FDG avidity ("signature" for FDG avidity) | 2 years
Differences in molecular and genetic profiles between FDG-positive polyps and FDG-positive cancers to suggest what gene mutations and abnormal mRNA and/or protein expressions may be required for cancer formation ("signature" for cancer) | 2 years
Differences in molecular and genetic profiles between normal colonic mucosa, polyps, and cancer | 2 years
Differences and similarities in molecular and genetic profiles between FDG-positive cancers and polyps | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marc J. Gollub, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Suresh Jhanwar, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States